CLINICAL TRIAL: NCT05382364
Title: A Phase 1 Clinical Study to Investigate the Safety and Pharmacokinetics of Tucatinib (MK-7119) in China Participants With HER2+ Advanced Breast Cancer, Gastric or Gastroesophageal Junction Adenocarcinoma and Colorectal Cancer
Brief Title: Safety and Pharmacokinetics of Tucatinib (MK-7119) in Chinese Participants With Cancer (MK-7119-002)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-7119-002; C4251016 (Other: Alias Study Number); 7119-002 (Other: Alias Study Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Metastatic HER2+ Advanced Breast Cancer; Breast Neoplasms; Gastric or Gastroesophageal Junction Adenocarcinoma (GEC); Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — tucatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tucatinib Treatment (Experimental): Chinese participants with HER2+ advanced breast cancer, gastric or gastroesophageal junction adenocarcinoma, or colorectal cancer receive tucatinib 300 mg by mouth twice daily during 21-day cycles. Treatment continues until there is evidence of unacceptable toxicity or documented progression.
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Tucatinib — Tucatinib 150 mg and 50 mg tablets taken by mouth at a dose of 300 mg twice daily.
  Other Names: MK-7119

SUMMARY:
The primary purpose of this study is to characterize the safety and tolerability of tucatinib (MK-7119) in Chinese participants with human epidermal growth factor receptor 2 positive (HER2+) advanced breast cancer, gastric or gastroesophageal junction adenocarcinoma (GEC), and colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2+ advanced breast cancer, gastric or GEC, and colorectal cancer
* Have progressed at least one previous therapeutic regimen and either no longer are candidates for standard therapy, have no standard therapy available, or choose not to pursue standard therapy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance within 7 days prior to allocation
* Has life expectancy >6 months in the opinion of the investigator
* Have measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 as assessed by the local site investigator/radiologist
* Must test negative for hepatitis B surface antigen (HBsAg)
* If there is a history of hepatitis C virus (HCV) infection, has undetectable HCV viral load at screening
* For males, agree to be abstinent from heterosexual intercourse, or agree to use acceptable contraception, for the duration of study and 1 week after
* For females, is not pregnant or breastfeeding AND one of the following applies:
* Is not a woman of childbearing potential (WOCBP)
* Is a WOCBP and uses highly effective contraception and is not pregnant

Exclusion Criteria:

* History of prior cancer within <3 year, except for adequately treated basal cell or squamous cell carcinoma of the skin, cervical cancer in situ, or other in situ carcinomas which needs discussion between the investigator and the Sponsor
* Participants with leptomeningeal disease are excluded
* Has symptomatic central nervous system (CNS) metastases
* Has active human immunodeficiency virus (HIV), hepatitis B virus, or HCV infection
* Has had chemotherapy, immunotherapy, radioimmunotherapy, definitive radiation, or biological cancer therapy or treatment with an investigational product within 4 weeks (2 weeks for palliative radiation) before the first dose of study intervention
* Has an active infection requiring therapy
* Has refractory nausea/vomiting, chronic gastrointestinal disease, or significant bowel resection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study
* Has a QTc prolongation
* Has uncontrolled illness including but not limited to ongoing symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements
* Has had major surgery within 4 weeks prior to first dose of study intervention
* Is currently participating in another clinical trial
* Has psychiatric or substance abuse disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with ≥1 adverse event (AE) | Up to approximately 2.5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study therapy due to AE | Up to approximately 2.5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Cmax of tucatinib will be determined after the first dose.
Time of maximum plasma concentration (Tmax) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Tmax of tucatinib will be determined after the first dose.
Area under the plasma concentration time curve from dosing to 12 hours postdose (AUC0-12) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The AUC0-12 of tucatinib will be determined after the first dose.
Apparent plasma half-life (t½) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The t½ of tucatinib will be determined after the first dose.
Apparent clearance (CL/F) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The CL/F of tucatinib will be determined after the first dose.
Volume of distribution (Vz/F) of first dose of tucatinib | Cycle 1, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Vz/F of tucatinib will be determined after the first dose.
Trough concentration (Ctrough) of tucatinib at steady state | Cycle 1, Days 8 and 15: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Ctrough of tucatinib will be determined at steady state.
Accumulation ratio of tucatinib at steady state | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The accumulation ratio of tucatinib will be determined at steady state.
Cmax at steady state (Cmaxss) of tucatinib | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Cmaxss of tucatinib will be determined at steady state.
Tmax at steady state (Tmaxss) of tucatinib | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Tmaxss of tucatinib will be determined at steady state.
AUC0-12 at steady state (AUC0-12ss) of tucatinib | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The AUC0-12ss of tucatinib will be determined at steady state.
t½ of tucatinib at steady state | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The t½ of tucatinib will be determined at steady state.
CL/F at steady state (CL/Fss) of tucatinib | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The CL/Fss of tucatinib will be determined at steady state.
Vz/F at steady state (Vz/Fss) of tucatinib | Cycle 2, Day 1: predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose
  The Vz/Fss of tucatinib will be determined at steady state.
Objective Response Rate (ORR) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 19 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR based on RECIST 1.1 will be presented.
Duration of Response (DOR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 19 months
  For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- China (5):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MK-7119-002